CLINICAL TRIAL: NCT04076059
Title: China ARCHES: A Multicenter, Phase 3, Randomized, Double-blind, Placebo Controlled Efficacy and Safety Study of Enzalutamide Plus Androgen Deprivation Therapy (ADT) Versus Placebo Plus ADT in Chinese Patients With Metastatic Hormone Sensitive Prostate Cancer (mHSPC)
Brief Title: An Efficacy and Safety Study of Enzalutamide Plus Androgen Deprivation Therapy (ADT) Versus Placebo Plus ADT in Chinese Patients With Metastatic Hormone Sensitive Prostate Cancer (mHSPC)
Acronym: China ARCHES
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9785-CL-0336; CTR20190132 (Registry Identifier: ChinaDrugTrials.org.cn)
Record Dates: First submitted 2019-08-19; First posted 2019-09-03 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Hormone Sensitive Prostate Cancer
Keywords: Metastatic hormone sensitive prostate cancer; Androgen Deprivation Therapy (ADT); Xtandi; MDV3100; Enzalutamide
MeSH Terms: interventions — enzalutamide; Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) (Experimental): Participants received enzalutamide 160 mg capsules, orally once daily if tolerable, and continued ADT until radiographic disease progression was documented or until they started another investigational agent or new therapy for treatment of prostate cancer. Participants were to remain on study treatment until confirmed radiographic disease progression. ADT (either bilateral orchiectomy or LHRH agonist/antagonist) was maintained during study treatment.
  Interventions: Drug: Enzalutamide; Drug: Androgen deprivation therapy (ADT)
- Placebo Plus ADT (Double Blind Phase) (Placebo Comparator): Participants received enzalutamide-matching placebo capsules, orally once daily and continued ADT until radiographic disease progression was documented or until they started another investigational agent or new therapy for treatment of prostate cancer. Participants were to remain on study treatment until confirmed radiographic disease progression. ADT (either bilateral orchiectomy or LHRH agonist/antagonist) was maintained during study treatment."
  Interventions: Drug: Placebo; Drug: Androgen deprivation therapy (ADT)
- Enzalutamide Plus ADT (Open-Label Phase) (Experimental): Participants who received placebo in double-blind phase and remaind on study treatment until confirmed radiographic disease progression received enzalutamide and continued ADT in open-label phase. ADT (either bilateral orchiectomy or LHRH agonist/antagonist) was maintained during study treatment.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Oral
  Other Names: Xtandi; MDV3100
  Arms: Enzalutamide Plus ADT (Open-Label Phase); Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase)
Drug: Placebo — Oral
  Arms: Placebo Plus ADT (Double Blind Phase)
Drug: Androgen deprivation therapy (ADT) — All participants were required to maintain ADT during study treatment, either using luteinizing hormone-releasing hormone (LHRH) agonist/antagonist or having a history of bilateral orchiectomy.
  Arms: Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase); Placebo Plus ADT (Double Blind Phase)

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of enzalutamide plus androgen deprivation therapy (ADT) versus placebo plus ADT in Chinese subjects with metastatic hormone sensitive prostate cancer (mHSPC). The study was conducted in two phases: Double-Blind treatment phase and open-label phase.

ELIGIBILITY:
Inclusion Criteria:

Double Blind treatment Phase:

* Subject is diagnosed with histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation, signet cell or small cell histology.
* Subject has metastatic prostate cancer documented by positive bone scan (for bone disease) or measurable metastatic lesions on computed tomography (CT) or magnetic resonance imaging (MRI) scan (for soft tissue). Subjects whose disease spread is limited to regional pelvic lymph nodes are not eligible.
* Once randomized at day 1, subject must maintain androgen deprivation therapy (ADT) with a luteinizing hormone-releasing hormone (LHRH) agonist or antagonist during study treatment or have a history of bilateral orchiectomy (i.e., medical or surgical castration).
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening.
* Subject has an estimated life expectancy of ≥ 12 months.
* Subject is able to swallow the study drug and comply with study requirements.
* A sexually active male subject with female partner(s) who is of childbearing potential is eligible if:

  * Agrees to use a male condom starting at screening and continue throughout the study treatment and for at least 3 months after the last dose of study drug. If the male subject has not had a vasectomy or is not sterile at least 6 months prior to screening his female partner(s) is utilizing 1 form of highly effective birth control per locally accepted standards starting at screening and continue throughout study treatment and for at least 3 months after the male subject receives his last dose of study drug.
* Subject must agree to abstinence or use a condom throughout the study period and for at least 3 months after the last dose of study drug if engaging in sexual intercourse with a pregnant or breastfeeding partner(s).
* Subject must agree not to donate sperm from first dose of study drug through 3 months after the last dose of study drug.
* Subject agrees not to participate in another interventional study while on treatment.

Open Label Phase:

* Before the sponsor's formal determination on study-wide unblinding, includes the subject who has evidence of radiographic progression as confirmed during the double-blind treatment (only apply to the subject in the placebo arm).
* Subject has not met any of the discontinuation criteria in the main protocol. Subject in the placebo arm who achieved confirmed radiographic progression in the double-blinded period is eligible.
* Subject is willing to maintain ADT with LHRH agonist or antagonist or has had a bilateral orchiectomy
* Subject is able to swallow enzalutamide capsules whole and to comply with study requirements throughout the study
* Subject and subject's female partner agree to follow contraception and sperm donation requirements in main protocol
* IRB-/IEC-approved written informed consent and privacy language as per national regulations must be obtained from the subject or legally authorized representative prior to any study-related procedures (including withdrawal of prohibited medication, if applicable).
* Subject is considered an adult according to local regulation at the time of signing informed consent.
* After the sponsor's formal determination on study-wide unblinding, includes the subject who is randomized to receive treatment in the double-blind period (apply to all subjects).

Exclusion Criteria:

Double-Blind Treatment Phase:

* Subject has received any prior pharmacotherapy, radiation therapy or surgery for metastatic prostate cancer (the following exceptions are permitted):

  * Up to 3 months of ADT with LHRH agonists or antagonists or orchiectomy with or without concurrent antiandrogens prior to day 1, with no radiographic evidence of disease progression or rising prostate-specific antigen (PSA) levels prior to day 1;
  * Subject may have 1 course of palliative radiation or surgical therapy to treat symptoms resulting from metastatic disease if it was administered at least 4 weeks prior to day 1;
  * Up to 6 cycles of docetaxel therapy with final treatment administration completed within 2 months of day 1 and no evidence of disease progression during or after the completion of docetaxel therapy;
  * Up to 6 months of ADT with LHRH agonists or antagonists or orchiectomy with or without concurrent antiandrogens prior to day 1 if subject was treated with docetaxel, with no radiographic evidence of disease progression or rising PSA levels prior to day 1;
  * Prior ADT given for < 39 months in duration and > 9 months before randomization as neoadjuvant/adjuvant therapy.
* Subject had a major surgery within 4 weeks prior to day 1.
* Subject received treatment with 5-α reductase inhibitors (finasteride, dutasteride) within 4 weeks prior to day 1.
* Subject received treatment with estrogens, cyprotoerone acetate or androgens within 4 weeks prior to day 1.
* Subject received treatment with systemic glucocorticoids greater than the equivalent of 10 mg per day of prednisone within 4 weeks prior to day 1, intended for the treatment of prostate cancer.
* Subject received treatment with herbal medications that have known hormonal antiprostate cancer activity and/or are known to decrease PSA levels within 4 weeks prior to day 1.
* Subject received prior aminoglutethimide, ketoconazole, abiraterone acetate or enzalutamide for the treatment of prostate cancer or participation in a clinical study of an investigational agent that inhibits the androgen receptor or androgen synthesis (e.g., TAK-700, ARN-509, ODM-201).
* Subject received investigational agent within 4 weeks prior to day 1.
* Subject has known or suspected brain metastasis or active leptomeningeal disease.
* Subject has a history of another invasive cancer within 3 years of screening, with the exception of fully treated cancers with a remote probability of recurrence.
* Subject has absolute neutrophil count < 1500/μL, platelet count < 100000/μL or hemoglobin < 10 g/dL (6.2 mmol/L) at screening. NOTE: May not have received any growth factors within 7 days or blood transfusions within 28 days prior to the hematology values obtained at screening.
* Subject has total bilirubin ≥ 1.5 x the upper limit of normal (except subjects with documented Gilbert's disease), or alanine aminotransferase or aspartate aminotransferase ≥ 2.5 x the upper limit of normal at screening.
* Subject has creatinine > 2 mg/dL (177 μmol/L) at screening.
* Subject has albumin < 3.0 g/dL (30 g/L) at screening.
* Subject has a history of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma, brain arteriovenous malformation).
* Subject has history of loss of consciousness or transient ischemic attack within 12 months prior to day 1.
* Subject has clinically significant cardiovascular disease, including the following:

  * Myocardial infarction within 6 months prior to screening;
  * Unstable angina within 3 months prior to screening;
  * New York Heart Association class III or IV congestive heart failure or a history of New York Heart Association class III or IV congestive heart failure unless a screening echocardiogram or multigated acquisition scan performed within 3 months before the randomization date demonstrates a left ventricular ejection fraction ≥ 45%;
  * History of clinically significant ventricular arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes);
  * History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place;
  * Hypotension as indicated by systolic blood pressure < 86 mm Hg at screening;
  * Bradycardia as indicated by a heart rate of ≤ 45 beats per minute on the screening electrocardiogram;
  * Uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure measurements showing systolic blood pressure > 170 mm Hg or diastolic blood pressure > 105 mm Hg at screening.
* Subject has gastrointestinal disorder affecting absorption.
* Subject has any concurrent disease, infection or comorbid condition that interferes with the ability of the subject to participate in the study, which places the subject at undue risk or complicates the interpretation of data.
* Subject received bisphosphonates or denosumab within 2 weeks prior to day 1 unless administered at stable dose or to treat diagnosed osteoporosis.
* Subject has shown a hypersensitivity reaction to the active pharmaceutical ingredient or any of the study capsule components.

Open-Label Phase:

* Subject has taken commercially available enzalutamide
* After unblinding, subject has started any new investigational agent or anti-neoplastic therapy intended to treat prostate cancer
* Subject has any clinically significant disorder or condition including excessive alcohol or drug abuse, or secondary malignancy, which may interfere with study participation in the opinion of the investigator or medical monitor
* Subject has current or previously treated brain metastasis or active leptomeningeal disease
* Subject has a history of seizure or any condition that may increase the risk of seizure
* Subject's disease has progressed radiographically during the double-blind period of the study and treatment with study drug was stopped prior to study-wide unblinding. (Note: Subject who progressed radiographically while in the double-blind period of the study and continued treatment per protocol is allowed to participate in the open-label phase.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2028-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Science Manager, Study Director — Astellas Pharma China, Inc.
Locations (28):
- China (28):
  - Site CN86022, Beijing
  - Site CN86035, Beijing
  - Site CN86024, Changchun
  - Site CN86009, Changsha
  - Site CN86016, Changsha
  - Site CN86023, Changsha
  - Site CN86025, Fuzhou
  - Site CN86001, Guangzhou
  - Site CN86028, Hangzhou
  - Site CN86036, Hangzhou
  - Site CN86004, Nanchang
  - Site CN86002, Shanghai
  - Site CN86003, Shanghai
  - Site CN86010, Shanghai
  - Site CN86013, Shanghai
  - Site CN86014, Shanghai
  - Site CN86027, Shanghai
  - Site CN86020, Shenyang
  - Site CN86011, Shenzhen
  - Site CN86032, Suzhou
  - Site CN86012, Tianjin
  - Site CN86005, Ürümqi
  - Site CN86019, Wuhan
  - Site CN86026, Wuhan
  - Site CN86021, Wuxi
  - Site CN86038, Xi'an
  - Site CN86017, Zhengzhou
  - Site CN86029, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chinese men with metastatic hormone sensitive prostate cancer were enrolled in the study.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study. Randomization was stratified by volume of disease (low versus high) and prior docetaxel therapy for prostate cancer (no prior docetaxel, prior docetaxel).
Groups:
- Placebo Plus ADT (Double Blind Phase): Participants received enzalutamide-matching placebo capsules, orally once daily and continued ADT until radiographic disease progression was documented or until they started another investigational agent or new therapy for treatment of prostate cancer. Participants were to remain on study treatment until confirmed radiographic disease progression. ADT (either bilateral orchiectomy or LHRH agonist/antagonist) was maintained during study treatment.
Period: Double Blind Phase
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase) | Enzalutamide Plus ADT (Open-Label Phase)
Started | 120 | 60 | 0
Ongoing Participants | 82 | 18 | 0
Participants Who Received at Least One Dose of Study Drug | 119 | 59 | 0
Completed | 0 | 0 | 0
Not Completed | 120 | 60 | 0
Not completed — Progressive disease | 22 | 26 | 0
Not completed — Withdrawal by Subject | 4 | 11 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 5 | 1 | 0
Not completed — Ongoing Participants | 82 | 18 | 0
Not completed — Miscellaneous | 3 | 1 | 0
Not completed — Protocol Deviation | 1 | 1 | 0
Not completed — Did not take study drug | 1 | 1 | 0
Period: Open Label Phase
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase) | Enzalutamide Plus ADT (Open-Label Phase)
Started | 0 (Only participants who received placebo in the double blind Phase received enzalutamide plus ADT in Open -label Phase.) | 0 (Only participants who received placebo in the double blind Phase received enzalutamide plus ADT in Open -label Phase.) | 23 (Eligible participants who provided consent took part in open-label period)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 23
Not completed — Progressive disease | 0 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Death | 0 | 0 | 2
Not completed — Ongoing Participants | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase) | Total
Number analyzed (Participants) | 120 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.8 (7.4) | 68.7 (7.3) | 68.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 120 | 60 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 120 | 60 | 180
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 120 | 60 | 180
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Prior Docetaxel Use (yes or no) [Count of Participants; unit: Participants]
  Yes | 14 | 8 | 22
  No | 106 | 52 | 158
Volume of Disease (Low Vs High) [Count of Participants; unit: Participants]
  Low | 26 | 14 | 40
  High | 94 | 46 | 140

OUTCOME MEASURES:

1. Primary Outcome: Time to Prostrate Specific Antigen (PSA) Progression
Description: Time to PSA progression was calculated as the time from the date of randomization to the first observation of PSA progression. PSA progression was defined as a ≥ 25% increase and an absolute increase of ≥ 2 microgram/liter (μg/L) (2 nanogram/milliliter [ng/mL]) above the nadir (i.e., lowest PSA value observed post baseline or at baseline), which was confirmed by a second consecutive value at least 3 weeks later. Time to event analysis was performed using Kaplan-Meier estimates.
Time Frame: From the date of randomization to the first observation of PSA progression (up to 38 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase)
Number analyzed (Participants) | 120 | 60
Months | NA [NA to NA] — Not Reached. Data was not estimable due to low number of events | 9.2 [6.54 to 17.48]
Statistical Analysis 1: Comparison: Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) vs Placebo Plus ADT (Double Blind Phase); Test type: Superiority; p < 0.0001, Log Rank; Cox Proportional Hazard = 0.130, 95% CI 2-sided [0.076 to 0.222] — Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period

2. Secondary Outcome: Radiographic Progression-Free Survival (rPFS)
Description: An rPFS event was defined as the time from randomization to the first objective evidence of radiographic disease progression assessed by investigator or death (defined as death from any cause within 24 weeks from study drug discontinuation), whichever occurred first. Radiographic disease progression was defined as progressive disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for soft tissue disease or by appearance of 2 or more new lesions on bone scan. Time to event analysis was performed using Kaplan-Meier estimates.
Time Frame: up to 38 months
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase)
Number analyzed (Participants) | 120 | 60
Months | NA [28.25 to NA] — Not Reached. Median and upper CI was not estimable due to low number of events | 19.4 [13.63 to NA] — Not Reached. Upper CI was not estimable due to low number of events
Statistical Analysis 1: Comparison: Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) vs Placebo Plus ADT (Double Blind Phase); Test type: Superiority; p < 0.0001, Log Rank; Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period; Cox Proportional Hazard = 0.330, 95% CI 2-sided [0.196 to 0.556]

3. Secondary Outcome: Time to First Symptomatic Skeletal Event (SSE)
Description: Time to first SSE was defined as the time from randomization to the occurrence of the first SSE. SSE was defined as radiation or surgery to bone, clinically apparent pathological bone fracture or spinal cord compression. Time to event analysis was performed using Kaplan-Meier estimates.
Time Frame: Up to 38 months
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase)
Number analyzed (Participants) | 120 | 60
Months | NA [NA to NA] — Not Reached. Data was not reached due to low number of events | NA [NA to NA] — Not Reached. Data was not reached due to low number of events
Statistical Analysis 1: Comparison: Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) vs Placebo Plus ADT (Double Blind Phase); Test type: Superiority; p = 0.7279, Log Rank; Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period; Cox Proportional Hazard = 0.789, 95% CI 2-sided [0.208 to 2.998]

4. Secondary Outcome: Time to Castration Resistance
Description: Castration resistance was defined as occurrence of radiographic disease progression, PSA progression or SSE with castrate levels of testosterone (< 50 ng/dL). Time to castration resistance was defined as the time from randomization to the first castration resistant event (radiographic disease progression, PSA progression or SSE), whichever occurred first. PSA progression was defined as a ≥ 25% increase and an absolute increase of ≥ 2 μg/L (2 ng/mL) above the nadir (i.e., lowest PSA value observed post baseline or at baseline), which was confirmed by a second consecutive value at least 3 weeks later. Radiographic disease progression was defined as progressive disease by RECIST version 1.1 for soft tissue disease or by appearance of 2 or more new lesions on bone scan. SSE was defined as radiation or surgery to bone, clinically apparent pathological bone fracture or spinal cord compression. Time to event analysis was performed using Kaplan-Meier estimates.
Time Frame: Up to 38 months
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase)
Number analyzed (Participants) | 120 | 60
Months | NA [31.18 to NA] — Median and upper CI was not estimable due to low number of events | 8.3 [6.41 to 14.69]
Statistical Analysis 1: Comparison: Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) vs Placebo Plus ADT (Double Blind Phase); Test type: Superiority; p < 0.0001, Log Rank; Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period; Cox Proportional Hazard = 0.172, 95% CI 2-sided [0.107 to 0.276]

5. Secondary Outcome: Percentage of Participants With PSA Response (≥ 50%)
Description: The PSA response rate ≥50% is defined as the percentage of participants in the analysis population with maximal PSA declines of at least 50% at any time and at each visit for participants with detectable PSA at baseline and at least 1 post-baseline assessment.
Time Frame: Up to 38 months
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase)
Number analyzed (Participants) | 120 | 60
Percentage of participants | 93.3 [87.3 to 97.1] | 80.0 [67.7 to 89.2]
Statistical Analysis 1: Comparison: Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) vs Placebo Plus ADT (Double Blind Phase); Test type: Superiority; p = 0.0036, Cochran-Mantel-Haenszel; Stratified by volume of disease and previous docetaxel use during screening period. Parameter estimate: Difference in percentage

6. Secondary Outcome: Percentage of Participants With PSA Response (≥ 90%)
Description: The PSA response rate ≥90% is defined as the percentage of participants in the analysis population with maximal PSA declines of at least 90% at any time and at each visit for participants with detectable PSA at baseline and at least 1 post-baseline assessment.
Time Frame: Up to 38 months
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase)
Number analyzed (Participants) | 120 | 60
Percentage of participants | 86.7 [79.3 to 92.2] | 55.0 [41.6 to 67.9]
Statistical Analysis 1: Comparison: Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) vs Placebo Plus ADT (Double Blind Phase); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 5, analysis 1]

7. Secondary Outcome: Time to Initiation of New Antineoplastic Therapy
Description: Time to initiate of a new antineoplastic therapy (including cytotoxic and hormone therapies) was defined as the time interval from randomization to the date of the first dose administration of the first antineoplastic therapy. Time to event analysis was performed using Kaplan-Meier estimates.
Time Frame: Up to 38 months
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase)
Number analyzed (Participants) | 120 | 60
Months | NA [NA to NA] — Not Reached. Data was not reached due to low number of events | 31.1 [NA to NA] — Not Reached. Data was not reached due to low number of events
Statistical Analysis 1: Comparison: Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) vs Placebo Plus ADT (Double Blind Phase); Test type: Superiority; p = 0.5899, Log Rank; Stratified by volume of disease (low vs high) and prior docetaxel use (yes vs no) during screening period; Cox Proportional Hazard = 0.797, 95% CI 2-sided [0.350 to 1.819]

8. Secondary Outcome: Percentage of Participants With Undetectable PSA (< 0.2 ng/mL)
Description: The PSA undetectable rate was defined as the percentage of participants with detectable (≥ 0.2 ng/mL) PSA at baseline, which became undetectable (< 0.2 ng/mL) during study treatment. Only participants with detectable PSA at baseline was included in the analysis.
Time Frame: Up to 38 months
Population: ITT Population with detectable PSA at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase)
Number analyzed (Participants) | 114 | 57
Percentage of participants | 76.3 [67.4 to 83.8] | 22.8 [12.7 to 35.8]
Statistical Analysis 1: Comparison: Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) vs Placebo Plus ADT (Double Blind Phase); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 5, analysis 1]; Difference in Percentage = 53.5, 95% CI 2-sided [40.1 to 66.9]

9. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of participants with measurable disease at baseline who achieved a complete or partial response (CR or PR) in their soft tissue disease using the RECIST version 1.1 criteria, CR was defined as complete disappearance of all target lesions and non-target disease. No new lesions. PR was defined as >=30% decrease on study under baseline of the sum of longest diameters of all target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Up to 38 months
Population: ITT Population with measurable soft tissue disease at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase)
Number analyzed (Participants) | 47 | 22
Percentage of participants | 76.6 [62.0 to 87.7] | 81.8 [59.7 to 94.8]
Statistical Analysis 1: Comparison: Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) vs Placebo Plus ADT (Double Blind Phase); Test type: Superiority; p = 0.8312, Cochran-Mantel-Haenszel; [statistical method as in outcome 5, analysis 1]; Difference in Percentage = -5.2, 95% CI 2-sided [-25.4 to 14.9]

ADVERSE EVENTS:
Time Frame: From the first dose up to 38 months
Description: The safety (SAF) population included all randomized participants who received at least 1 dose of study drug. Data reported for deaths are the number of participants who died regardless of time (could be beyond treatment emergent adverse event time frame).
Arm/Group | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) | Placebo Plus ADT (Double Blind Phase) | Enzalutamide Plus ADT (Open-Label Phase)
All-Cause Mortality (participants affected / at risk) | 21/119 | 12/59 | 8/23
Serious Adverse Events (participants affected / at risk) | 42/119 | 12/59 | 5/23
Other Adverse Events (participants affected / at risk) | 115/119 | 54/59 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) (N=119) | Placebo Plus ADT (Double Blind Phase) (N=59) | Enzalutamide Plus ADT (Open-Label Phase) (N=23)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Mesenteric artery embolism (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (9) | 1 (2) | 0 (0)
Liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 1 (2)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 8 (10) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 0 (0) | 0 (0)
Penetrating aortic ulcer (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide Plus Androgen Deprivation Therapy (ADT) (Double Blind Phase) (N=119) | Placebo Plus ADT (Double Blind Phase) (N=59) | Enzalutamide Plus ADT (Open-Label Phase) (N=23)
Anaemia (Blood and lymphatic system disorders) | 41 (106) | 23 (45) | 6 (13)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 10 (11) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (10) | 3 (3) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 3 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (7) | 5 (5) | 0 (0)
Toothache (Gastrointestinal disorders) | 9 (9) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (7) | 1 (1) | 1 (1)
Asthenia (General disorders) | 7 (7) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 3 (7) | 0 (0)
Fatigue (General disorders) | 18 (21) | 6 (7) | 2 (2)
Malaise (General disorders) | 11 (11) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 14 (20) | 4 (5) | 0 (0)
Pyrexia (General disorders) | 4 (6) | 3 (4) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (5) | 3 (5) | 0 (0)
Mastoiditis (Infections and infestations) | 10 (11) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 8 (8) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (15) | 5 (6) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 6 (8) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 22 (52) | 15 (32) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 23 (32) | 13 (25) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 9 (28) | 11 (26) | 4 (6)
Blood bilirubin increased (Investigations) | 13 (33) | 9 (16) | 1 (1)
Blood creatinine increased (Investigations) | 7 (18) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 6 (7) | 4 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 8 (60) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 7 (25) | 3 (8) | 2 (5)
Weight decreased (Investigations) | 11 (20) | 5 (7) | 2 (2)
Weight increased (Investigations) | 50 (208) | 19 (46) | 4 (6)
White blood cell count decreased (Investigations) | 8 (58) | 2 (13) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 19 (22) | 5 (8) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 12 (33) | 3 (6) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 14 (36) | 8 (18) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 31 (89) | 12 (32) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (5) | 4 (6) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 12 (28) | 4 (10) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 (6) | 5 (6) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 10 (32) | 4 (6) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 33 (147) | 12 (42) | 3 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 15 (41) | 7 (16) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (13) | 5 (7) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 8 (24) | 6 (8) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (28) | 9 (21) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (11) | 6 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (23) | 9 (10) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 7 (10) | 2 (2) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (25) | 3 (4) | 3 (4)
Bone hypertrophy (Musculoskeletal and connective tissue disorders) | 10 (40) | 0 (0) | 2 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (18) | 12 (16) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 1 (1) | 2 (4)
Osteitis (Musculoskeletal and connective tissue disorders) | 14 (29) | 1 (2) | 3 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (11) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (17) | 5 (8) | 0 (0)
Dizziness (Nervous system disorders) | 15 (19) | 8 (11) | 1 (1)
Headache (Nervous system disorders) | 9 (9) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 10 (13) | 3 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 15 (18) | 3 (4) | 0 (0)
Dysuria (Renal and urinary disorders) | 10 (16) | 2 (5) | 1 (1)
Haematuria (Renal and urinary disorders) | 9 (23) | 3 (6) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 9 (10) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 11 (14) | 6 (7) | 1 (1)
Urinary retention (Renal and urinary disorders) | 5 (6) | 4 (4) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 23 (28) | 9 (9) | 2 (2)
Hypertension (Vascular disorders) | 30 (68) | 19 (41) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators (PI) are NOT employed by the organization sponsoring the study. There IS an agreement between PI's and the Sponsor that restricts the PI's rights to discuss or publish trial results after the trial is completed. Institute and/or PI may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT04076059/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT04076059/SAP_001.pdf